CLINICAL TRIAL: NCT05349305
Title: Population Pharmacokinetics and Individualized Administration of Lassila Tazobactam in Patients Undergoing CRRT After Aortic Dissection
Brief Title: Population Pharmacokinetics of Lassila Tazobactam in Patients After Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: byssc1985
Record Dates: First submitted 2022-04-19; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Aortic Dissection; Lung Infection
Keywords: Piperacillin tazobactam; CRRT
MeSH Terms: conditions — Aortic Dissection | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: continuous renal replacement therapy — continuous renal replacement therapy
  Other Names: non

SUMMARY:
The individualized drug use research on optimizing piperacillin tazobactam for CRRT of hospital-acquired pulmonary infection after cardiopulmonary bypass is still in the initial stage at home and abroad, lacking systematic research data. With the help of the population pharmacokinetic model, it can help clinicians to formulate individualized drug administration plans for such patients and provide methodological and data support for precise treatment. The rational use of piperacillin tazobactam will play an important role in reducing the use of carbapenems and curbing the occurrence of drug resistance.

DETAILED DESCRIPTION:
The incidence of acute renal failure after aortic dissection can be as high as 30%. In order to reduce mortality, most patients need continuous renal replacement therapy (CRRT). The concentration of antimicrobial drugs in patients receiving CRRT is often lower than the treatment level, which leads to treatment failure. The drug clearance rate of critically ill patients may change every day and it is difficult to estimate, especially when the renal function deteriorates and CRRT begins.

As a time-dependent antimicrobial drug, increasing the% t > MIC of piperacillin tazobactam is closely related to ensuring clinical efficacy. However, the molecular weight of piperacillin tazobactam is less than 2000 d, which can easily pass through the filter membrane. All CRRT methods have the same clearance rate. Meanwhile, the binding rate of piperacillin and tazobactam to plasma protein is only about 30%, which is easy to clear through CRRT. As a result, the curative effect of piperacillin tazobactam in treating hospital-acquired pneumonia after aortic dissection is not good according to the conventional dosage and administration. More and more doctors will consider choosing carbapenems as soon as possible, which is related to national health.

Therefore, the traditional pharmacokinetic study is no longer applicable, and it can't provide a basis for clinical determination of individualized drug use plan of piperacillin and tazobactam, while the population pharmacokinetic study can effectively solve this problem. The frequency of blood collection from patients is low (usually 2 ~ 4 blood collection points), which is the most advanced method for individualized drug use research in the world at present [10]. Methods The Nonlinear mixed effect Model (non-MEM) was used to calculate the average and variability of pharmacokinetic parameters in patients, and the synergistic effect of patient factors (such as age and weight) on pharmacokinetic parameters could be evaluated, thus providing a reliable basis for formulating individualized and accurate drug administration plan and improving the success rate of anti-infection.

ELIGIBILITY:
Inclusion Criteria:

Cardiopulmonary bypass during aortic dissection， Lung infection， Continuous renal replacement therapy

Exclusion Criteria:

Intracranial infection, Urinary tract infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with pulmonary infection after aortic dissection treated with CRRT and piperacillin tazobactam
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
blood concentration | Up to 8 hours after administration
  Blood concentration of piperacillin and tazobactam in whole period after administration

IPD SHARING:
Plan to Share IPD: Undecided